CLINICAL TRIAL: NCT01975610
Title: A Phase 2a, 4-Week Double-Blind, Proof-of-Concept Efficacy and Safety Study of CC-292 Versus Placebo as Co-therapy With Methotrexate in Active Rheumatoid Arthritis
Brief Title: Efficacy and Safety Study of CC-292 Versus Placebo as Co-therapy With Methotrexate in Active Rheumatoid Arthritis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CC-292-RA-001
Record Dates: First submitted 2013-10-29; First posted 2013-11-04 (Estimated); Last update posted 2017-07-31 (Actual); Status verified 2017-07

CONDITIONS: Rheumatoid Arthritis
Keywords: Arthritis, Rheumatoid, Autoimmune, Inflammatory, Synovial, Bruton's tyrosine kinase (Btk), CC-292, Joint Disease
MeSH Terms: conditions — Arthritis, Rheumatoid; Arthritis; Joint Diseases | interventions — spebrutinib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- CC-292 375mg (Experimental): Treatment
  Interventions: Drug: CC-292
- Placebo (Placebo Comparator): Control
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: CC-292 — 375 mg PO daily (250 mg in the AM and 125 mg in the PM for 28 days)
  Arms: CC-292 375mg
Drug: Placebo — Twice daily for 28 days
  Arms: Placebo

SUMMARY:
CC-292 is an oral agent that is under clinical development for the treatment of rheumatoid arthritis an autoimmune inflammatory disorder.

This study will test the clinical effectiveness and safety of an orally (PO) administered dose of CC-292 compared to placebo in US female patients currently on background Methotrexate (MTX) with active Rheumatoid Arthritis (RA

DETAILED DESCRIPTION:
This is a Phase 2a, multicenter, randomized, double-blind, placebo-controlled, proof-of-concept study to determine the efficacy and safety of CC-292 (375 mg PO daily) on a stable background of MTX therapy in female subjects with active RA.

Approximately 80 female subjects with active RA will be randomized 1:1 into two dose groups: active CC-292 (375 mg PO daily) or identically-appearing placebo capsules for 4 weeks

ELIGIBILITY:
Inclusion Criteria:

* Female between 18 and 80 years of age (inclusive) at the time of signing the informed consent.
* Must meet the 2010 ACR/EULAR Classification Criteria for RA (Appendix A), have RA for at least 6 months and must continue to have active RA at the time of randomization despite at least 3 months of treatment with stable doses of MTX (7.5 to 25 mg/week oral or parenteral) for at least 4 weeks prior to randomization.
* Must have been treated with MTX for at least 3 months prior to randomization, and must be on a stable dose between 7.5 and 25 mg/week (PO or parenteral, not both) for at least 4 weeks prior to randomization. Subjects will be required to maintain their stable dose through Day 28/Week 4 of the study. Oral folate supplementation is required with a minimum dose of 5 mg/week (ie, folic acid) while the subject is taking MTX. Leucovorin may be used instead of folic acid and may be dosed up to 10 mg/week orally.
* Sulfasalazine is allowed as a concomitant medication, however, subject must be on a stable dose for at least 4 weeks prior to randomization and through Day 28/Week 4 of the study.
* Hydroxychloroquine or chloroquine is allowed as concomitant medications, however, subject must be on a stable dose for at least 4 weeks prior to randomization and through Day 28/Week 4 of the study.
* Modification of Diet in Renal Disease formula (MDRD) estimated glomerular filtration rate (MDRD eGFR) ≥ 60 mL/min/1.73m2+

Exclusion Criteria:

* Male subjects
* Any condition that could affect CC-292 absorption, including gastric restrictions, bariatric surgery, such as gastric bypass, and clinical conditions that are associated with decreased intragastric acid production such as acid pernicious anemia.
* Currently using treatment with DMARDs (other than sulfasalazine, hydroxychloroquine or chloroquine and MTX), including biologics. Previous use is only allowed after adequate washout (4 weeks or 5 half-lives, whichever is longer) prior to randomization.
* Previous treatment with any cell depleting therapies, including investigational agents (eg, CAMPATH, anti-CD4, anti-CD5, anti-CD3, anti-CD19 and anti-CD20) within 6 months of screening.
* Treatment with intravenous gamma globulin, plasmapheresis or Prosorba® column within 2 weeks prior to randomization.
* Intra-articular or parenteral corticosteroids are not allowed within 2 weeks prior to randomization.

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2013-10; Primary Completion 2016-01 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
American College of Rheumatology Criteria for a 20% improvement (ACR 20) | Week 4
  Percentage of participants with an American College of Rheumatology ≥20% (ACR20) response. A participant is a responder if the following 3 criteria for improvement from Baseline are met: • ≥ 20% improvement in 68 tender joint count; • ≥ 20% improvement in 66 swollen joint count; and • ≥ 20% improvement in at least 3 of the 5 following parameters: o Patient's assessment of pain (measured on a 100 mm visual analog scale [VAS]); o Patient's global assessment of disease activity (measured on a 100 mm VAS); o Physician's global assessment of disease activity (measured on a 100 mm VAS); o Patient's self-assessment of physical function (Health Assessment Questionnaire - Disability Index (HAQ-DI)); o C-Reactive Protein

SECONDARY OUTCOMES:
Number of participants with adverse events | Up to 8 Weeks
  Safety and tolerability of CC-292 compared with placebo in subjects on a background of stable MTX therapy. An adverse event (AE) is any noxious, unintended, or untoward medical occurrence that may appear or worsen in a subject during the course of a study. It may be a new intercurrent illness, a worsening concomitant illness, an injury, or any concomitant impairment of the subject's health, including laboratory test values (as specified by the criteria below), regardless of etiology. Any worsening (ie, any clinically significant adverse change in the frequency or intensity of a preexisting condition) should be considered an AE.
American College of Rheumatology Criteria for a 50% improvement (ACR 50) | Week 4
  Percentage of participants with an American College of Rheumatology ≥50% (ACR50) response. A participant is a responder if the following 3 criteria for improvement from Baseline are met:
  * ≥ 50% improvement in 68 tender joint count;
  * ≥ 50% improvement in 66 swollen joint count; and
  * ≥ 50% improvement in at least 3 of the 5 following parameters:
    * Patient's assessment of pain (measured on a 100 mm visual analog scale [VAS]);
    * Patient's global assessment of disease activity (measured on a 100 mm VAS);
    * Physician's global assessment of disease activity (measured on a 100 mm VAS);
    * Patient's self-assessment of physical function (Health Assessment Questionnaire - Disability Index (HAQ-DI));
    * C-Reactive Protein.
American College of Rheumatology Criteria for a 70% improvement (ACR 70) | Week 4
  Percentage of participants with an American College of Rheumatology ≥70% (ACR70) response. A participant is a responder if the following 3 criteria for improvement from Baseline are met:
  * ≥ 70% improvement in 68 tender joint count;
  * ≥ 70% improvement in 66 swollen joint count; and
  * ≥ 70% improvement in at least 3 of the 5 following parameters:
    * Patient's assessment of pain (measured on a 100 mm visual analog scale [VAS]);
    * Patient's global assessment of disease activity (measured on a 100 mm VAS);
    * Physician's global assessment of disease activity (measured on a 100 mm VAS);
    * Patient's self-assessment of physical function (Health Assessment Questionnaire - Disability Index (HAQ-DI));
    * C-Reactive Protein.

CONTACTS AND LOCATIONS:
Overall Officials: Douglas Hough, MD, MBA, Study Director — Celgene Corporation
Locations (27):
- United States (27):
  - Achieve Clinical Research LLC, Birmingham, Alabama
  - Arizona Arthritis and Rheumatology Research, PLLC, Phoenix, Arizona
  - Generations Medical Research, Hot Springs, Arkansas
  - UCLA, Los Angeles, California
  - Joao Nascimento, MD, Bridgeport, Connecticut
  - Southeastern Integrated Medical, Gainesville, Florida
  - Family Arthritis Center, Jupiter, Florida
  - Ocala Rheumatology Research Center, Ocala, Florida
  - Integral Rheumatology and Immunology specialists, Plantation, Florida
  - Columbia Medical Practice, Columbia, Maryland
  - Clinical Pharmacology Study Group, Worcester, Massachusetts
  - Borgess Research Institute, Kalamazoo, Michigan
  - Arthritis and Osteoporosis Associates, Freehold, New Jersey
  - Albuquerque Clinic, Albuquerque, New Mexico
  - NYU Langone Medical Center, New York, New York
  - DJL Clinical Research, Charlotte, North Carolina
  - Lynn Health Science Instiute, Oklahoma City, Oklahoma
  - Altoona Center for Clinical Research, Duncansville, Pennsylvania
  - Med Univ of South Carolina, Charleston, South Carolina
  - PMG Research of Charlotte LLC, Rock Hill, South Carolina
  - West Tennessee Research Institute, Jackson, Tennessee
  - Ramesh C Gupta MD, Memphis, Tennessee
  - Austin Regional Clinic, Austin, Texas
  - DM Clinical Research, Houston, Texas
  - Mountain State Clinical Research, Clarksburg, West Virginia
  - Froedtert Hospital BMT Medical College of Wisconsin, Milwaukee, Wisconsin
  - Gundersen Clinic Ltd, Onalaska, Wisconsin

REFERENCES:
- [Derived] Schafer PH, Kivitz AJ, Ma J, Korish S, Sutherland D, Li L, Azaryan A, Kosek J, Adams M, Capone L, Hur EM, Hough DR, Ringheim GE. Spebrutinib (CC-292) Affects Markers of B Cell Activation, Chemotaxis, and Osteoclasts in Patients with Rheumatoid Arthritis: Results from a Mechanistic Study. Rheumatol Ther. 2020 Mar;7(1):101-119. doi: 10.1007/s40744-019-00182-7. Epub 2019 Nov 13. PMID 31721017